CLINICAL TRIAL: NCT02407249
Title: Control for EU (European Union) Focal Impulse and Rotor Modulation Registry - Topera C-FIRM Registry-
Brief Title: Topera C-FIRM Registry
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Collaborators: I-Med-Pro GmbH (Other)
Responsible Party: Sponsor
Other Study IDs: C-FIRM-02
Record Dates: First submitted 2015-03-30; First posted 2015-04-02 (Estimated); Results first posted 2019-10-16 (Actual); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a control registry to the E-FIRM registry to track conventional atrial fibrillation (AF) procedures in terms of clinical usage, handling, and the safety and effectiveness for the treatment of symptomatic atrial fibrillation. Conventional AF ablation is defined as pulmonary vein isolation (PVI) and any additional ablation for AF according to the standard routine of the center.

Data items will be collected, if available, consistent and applicable with routine and standard clinical care at each participating site.

DETAILED DESCRIPTION:
Prospective and retrospective enrollment possible

ELIGIBILITY:
Inclusion Criteria:

* reported incidence of at least 2 documented episodes of symptomatic AF (paroxysmal, persistent or long standing persistent) during the 3 months preceding the initial AF ablation
* attempt of at least one Class I or III anti-arrhythmia drug with failure defined as recurrence of symptomatic AF or adverse drug effect resulting in stopping medication

Exclusion Criteria:

* women who are pregnant

As this is a registry only data of patients will be included who have been treated according to the current AF guidelines and the daily routine of the center.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Each participating site will enroll 10 consecutive conventional AF patients who are treated according to the standard routine of the center. Patients eligible should be in accordance with the AF Guidelines.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2015-04; Primary Completion 2017-05-31 (Actual); Study Completion 2018-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Hindricks, Prof. Dr., Principal Investigator — Herzzentrum Leipzig - Universitätsklinik; Kristin Ruffner, PhD, Study Director — Abbott
Locations (9):
- Germany (8):
  - Städtisches Klinikum Karlsruhe GmbH, Karlsruhe, Baden-Würtemberg
  - Herz- und Gefäßklinik, Bad Neustadt an der Saale, Bavaria
  - Klinikum Coburg GmbH, Coburg, Bavaria
  - Kardiologische Gemeinschaftspraxis am Park Sanssouci, Potsdam, Brandenburg
  - Herz- und Diabeteszentrum NRW, Bad Oeynhausen, North Rhine-Westphalia
  - Zentrum für klinische Prüfungen in der Facharztzentrum Dresden-Neustadt GbR, Dresden, Saxony
  - Herzzentrum Leipzig, Leipzig, Saxony
  - Unfallkrankenhaus Berlin, Berlin
- Erasmus Medical Center, Rotterdam, Netherlands

RESULTS

PARTICIPANT FLOW:
Groups:
- Registry Population: All participants enrolled in the C-FIRM registry.
Period: Overall Study
Arm/Group | Registry Population
Started | 73
Treated | 60
Completed | 47
Not Completed | 26
Not completed — Did not complete 12-month follow-up | 13
Not completed — Not treated | 13

BASELINE CHARACTERISTICS:
Population: Enrolled population
Arm/Group | Registry Population
Number analyzed (Participants) | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.2 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 53
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 29.0 (5.1)
New York Heart Association Class [Count of Participants; unit: Participants] — The New York Heart Association Functional Classification provides a simple way of classifying the extent of heart failure. It places patients in one of four categories based on how much they are limited during physical activity; the limitations/symptoms are in regard to normal breathing and varying degrees in shortness of breath and/or angina.
  Class I = no limitation of physical activity. Class II = slight limitation Class III = marked limitation Class IV = unable to carry on any physical activity without discomfort
  Participants
    Class I | 21
    Class II | 20
    Class III | 5
    Not reported | 27
Type of Atrial Fibrillation [Count of Participants; unit: Participants]
  Paroxysmal | 32
  Persistent | 40
  Not reported | 1
Left Ventricle Ejection Fraction [Mean (Standard Deviation); unit: percent] | 57.8 (9.0)
Left Atrium Diamter [Mean (Standard Deviation); unit: millimeter] | 45.2 (7.5)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Acute Success
Description: Acute Success was defined as elimination (by ablation) of pulmonary vein triggers during the procedure
Time Frame: day of procedure
Population: All treated patients
Measure: Count of Participants; unit: Participants
Groups:
- Analysis Population: All treated patients
Arm/Group | Analysis Population
Number analyzed (Participants) | 60
Participants | 53

2. Primary Outcome: Number of Participants With 12-Month Effectiveness
Description: Effectiveness success was defined as single procedure freedom from AF recurrence at 12-months after index procedure, excluding a 3-month blanking period.
Time Frame: 12 months after initial AF ablation
Population: Treated patients with 12-month follow-up data
Measure: Count of Participants; unit: Participants
Arm/Group | Analysis Population
Number analyzed (Participants) | 48
Participants | 34

3. Primary Outcome: Number of Participants With Acute Safety Success
Description: Acute safety success was defined as freedom from Serious Adverse Events 7 days after initial AF ablation
Time Frame: 7 days after initial AF ablation
Population: Analysis population for whom data are available
Measure: Count of Participants; unit: Participants
Arm/Group | Analysis Population
Number analyzed (Participants) | 57
Participants | 56

4. Primary Outcome: Number of Participants With 12-Month Safety Success
Description: 12-Month safety success was defined as freedom from Serious Averse Events at 12-months after index procedure
Time Frame: 12-months after index procedure
Population: Treated patients for whom 12-month safety data is available
Measure: Count of Participants; unit: Participants
Arm/Group | Analysis Population
Number analyzed (Participants) | 48
Participants | 45

5. Other Pre Specified Outcome: Number of Participants With 6-month Safety Success
Description: 6-Month safety success was defined as freedom from Serious Adverse Events 6-months after index procedure
Time Frame: 6-months after index procedure
Population: Treated patients for whom 6-month safety data is available
Measure: Count of Participants; unit: Participants
Arm/Group | Analysis Population
Number analyzed (Participants) | 54
Participants | 51

ADVERSE EVENTS:
Time Frame: 12-months
Groups:
- Enrolled Population: All patients enrolled in the registry
Arm/Group | Enrolled Population
All-Cause Mortality (participants affected / at risk) | 0/73
Serious Adverse Events (participants affected / at risk) | 3/73
Other Adverse Events (participants affected / at risk) | 0/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled Population (N=73)
Amaurosis fugax / volatile blindness right eye (Eye disorders) | 1 (1)
Strong hematoma left groin/knee (Vascular disorders) | 1 (1)
Ventricular extrasystole ablatiion (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Manuscripts prepared for publication will be submitted to sponsor for review and comments prior to submission to the publisher. This condition should not be construed as a means of restricting publication but is intended solely to assure mutual concurrence regarding data, evaluations, and conclusion, to provide an opportunity to share with the investigator any new and/or unpublished information of which he/she may be unaware, and to assure regulatory compliance of the results presented.

DOCUMENTS (1):
  • Study Protocol (2014-07-29): https://cdn.clinicaltrials.gov/large-docs/49/NCT02407249/Prot_000.pdf